CLINICAL TRIAL: NCT04154124
Title: Applying PET/MR in Rectal Cancer.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TASMC-19-ES-0448-CTIL
Record Dates: First submitted 2019-10-29; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rectal Cancer Patients (Experimental)
  Interventions: Diagnostic Test: PET/MR scan

INTERVENTIONS:
Diagnostic Test: PET/MR scan — whole-body PET/CT scan and pelvic PET/MR scan (MR protocol will include three plane fast spin echo T2 weighted, DWI and dynamic contrast enhanced imaging). The ad interim assessment will use a pelvic PET/MR scan only (without PET/CT), to avoid the radiation associated with whole body CT. In the staging and post-nT assessment, the addition of PET/MR to the standard use of PET/CT adds no radiation exposure.

SUMMARY:
The use of the novel recently introduced PET/MR scanner is believed to be promising in RC management, providing great anatomical details and detailed metabolic characterization. Preliminary data indicate it may become a strong imaging modality for staging of RC and has the potential to be used as a predictive tool guiding individualized therapy in patients receiving nT, but confirmation on prospective studies is mandatory. The use of radiomics as analysis approach may assist in achieving a better understanding of the obtained image data, and thus a more accurate disease assessment.

Objectives

1. To preliminary assess the potential diagnostic value of single PET/MR scan in RC staging and compare it to that of MRI alone, PET/CT alone, and combined MRI and PET/CT.
2. To preliminary assess the potential value of PET/MR in predicting pMR to nT.
3. To use radiomics analysis of PET/MR data to develop a quantification clinical tools that allow a more accurate and comprehensive assessment of RC patients.

ELIGIBILITY:
Inclusion Criteria:

1.Patients with newly diagnosed RC; histopathological confirmation of adenocarcinoma of colorectal origin.

Exclusion Criteria:

1. Patients younger than 18 years;
2. pregnancy;
3. other known active malignancy;
4. previous chemotherapy or radiotherapy;
5. previous pelvic operation;
6. patient that no intent / not suited for neoadjuvant therapy (including metastatic disease at presentation); contraindication to intravenous contrast agents.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-11-23 (Estimated); Primary Completion 2020-12-23 (Estimated); Study Completion 2021-12-23 (Estimated)

PRIMARY OUTCOMES:
Number of patient that shown the different between diagnostic value of single PET/MR scan in RC staging and compare it to that of MRI alone, PET/CT alone, and combined MRI and PET/CT | 1 year

IPD SHARING:
Plan to Share IPD: Undecided